CLINICAL TRIAL: NCT05885152
Title: Acute Effect of Whole-body Electrical Stimulation in COPD Patients: a Crossover Randomized Clinical Trial
Brief Title: Acute Effect of Whole-body Electrical Stimulation in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Jociane Schardong, Principal Investigator, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WBES_COPD
Record Dates: First submitted 2023-04-06; First posted 2023-06-01 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Whole-body electrical stimulation, Protocol 1 (Experimental): A whole body electrical stimulation session. Symmetrical biphasic current will be used, pulse width of 400µs, frequency of 75Hz, contraction time of five seconds, rest time of 10 seconds, for eight minutes, totaling 32 muscle contractions. During the first two minutes of stimulation, the patient will remain in isometry to become familiar with the electrical current. Then with the use of a stick (for proprioception), a series of biceps exercises and a series of triceps exercises, a series of sit-ups and a squat, a series of step ups and downs, and a series of plantings.
  Interventions: Other: Whole-body electrical stimulation
- Whole-body electrical stimulation, Protocol 2 (Experimental): A whole body electrical stimulation session. Symmetrical biphasic current will be used, pulse width of 400µs, frequency of 75Hz, contraction time of five seconds, rest time of 10 seconds, for 16 minutes, totaling 64 muscle contractions. During the first two minutes of stimulation, the patient will remain in isometry to become familiar with the electrical current. Then with the use of a stick (for proprioception), a series of biceps exercises and a series of triceps exercises, a series of sit-ups and a squat, a series of step ups and downs, and a series of plantings.
  Interventions: Other: Whole-body electrical stimulation

INTERVENTIONS:
Other: Whole-body electrical stimulation — Performed using Miha Bodytec equipment, properly calibrated, with electrodes on the quadriceps, hamstrings, glutes, biceps, triceps, pectorals, abdomen, trapezius, latissimus dorsi and quadratus lumborum muscles.
  Other Names: Whole-body electromyostimulation

SUMMARY:
Patients with chronic respiratory diseases present in addition to respiratory symptoms, peripheral muscle dysfunction, which contributes to functional impairment. The aim of the study is to investigate the safety of whole-body electrical stimulation in patients with chronic obstructive pulmonary disease (COPD). Patients will perform two whole body electrostimulation protocols, with an interval of one week between them. The primary outcome will be the safety of electrical stimulation through peripheral oxygen saturation, respiratory rate, systolic blood pressure, diastolic blood pressure, heart rate, dyspnea and fatigue (Borg subjective perceived exertion scale), autonomic control (rate variability cardiac arrest) and occurrence of adverse events. Secondary outcomes will be muscle damage assessed by serum creatine kinase level, muscle fatigue assessed by serum lactate level, delayed onset muscle soreness assessed by visual numerical scale, and peripheral muscle strength by dynamometry.

DETAILED DESCRIPTION:
Patients with COPD will be submitted to two whole body electrostimulation protocols, with an interval of one week between them. Miha Bodytec equipment will be properly calibrated, with electrodes on the quadriceps, hamstrings, glutes, biceps, triceps, pectorals, abdomen, trapezius, latissimus dorsi and quadratus lumborum muscles. Symmetric pulsed biphasic current will be used, pulse width of 400µs, frequency of 75Hz, contraction time of five seconds, rest time of 10 seconds. Protocol 1 will take eight minutes resulting in 32 muscle contractions, and protocol 2 will take 16 minutes resulting in 64 muscle contractions. Initially, patients will undergo an assessment of autonomic control. Then, blood collection will be performed, the serum lactate level will be checked and muscle strength will be measured. Verification of systolic blood pressure, diastolic blood pressure, peripheral oxygen saturation, heart rate, respiratory rate and perception of dyspnea and fatigue (BORG) will occur immediately before and after the whole body electrical stimulation session. During the protocol, peripheral oxygen saturation, heart rate, respiratory rate and BORG will be checked. After the session, the serum lactate level will be checked, a new blood collection will be performed and autonomic control and muscle strength will be reassessed. After 24, 48 and 72 hours, new blood samples will be collected and muscle pain will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD GOLD 3 and 4;
* Age between 18 and 80 years;
* Ability to ambulate.

Exclusion Criteria:

* Cognitive dysfunction that prevents assessments from being carried out, as well as inability to understand and sign the informed consent form (ICF);
* Intolerance to the electrostimulator and/or change in skin sensitivity;
* Patients with stroke sequelae;
* Recent acute myocardial infarction (two months);
* Uncontrolled hypertension;
* New York Heart Association grade IV heart failure or decompensated;
* Unstable angina or arrhythmia;
* Peripheral vascular changes in lower limbs such as deep vein thrombosis;
* Disabling osteoarticular or musculoskeletal disease;
* Uncontrolled diabetes (glycemia > 300mg/dL);
* Patients with cancer and/or undergoing cancer treatment;
* Patients with systemic lupus erythematosus or other autoimmune disease;
* Artificial cardiac pacemaker;
* Epilepsy;
* Hemophilia;
* Liver and kidney diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Peripheral oxygen saturation | Baseline
  Peripheral oxygen saturation will be assessed by pulse oximetry
Peripheral oxygen saturation | Protocol 1: minute four; Protocol 2: minute eight
  Peripheral oxygen saturation will be assessed by pulse oximetry
Peripheral oxygen saturation | Immediately after the session
  Peripheral oxygen saturation will be assessed by pulse oximetry
Respiratory rate | Baseline
  Respiratory rate will be assessed by respiratory rate count for one minute
Respiratory rate | Protocol 1: minute four; Protocol 2: minute eight
  Respiratory rate will be assessed by respiratory rate count for one minute
Respiratory rate | Immediately after the session
  Respiratory rate will be assessed by respiratory rate count for one minute
Heart rate | Baseline
  Heart rate will be assessed by pulse oximetry
Heart rate | Protocol 1: minute four; Protocol 2: minute eight
  Heart rate will be assessed by pulse oximetry
Heart rate | Immediately after the session
  Heart rate will be assessed by pulse oximetry
Systolic blood pressure | Baseline
  Systolic blood pressure will be assessed through sphygmomanometer
Systolic blood pressure | Immediately after the session
  Systolic blood pressure will be assessed through sphygmomanometer
Diastolic blood pressure | Baseline
  Diastolic blood pressure will be assessed through sphygmomanometer
Diastolic blood pressure | Immediately after the session
  Diastolic blood pressure will be assessed through sphygmomanometer
Dyspnea and Fatigue | Baseline
  Dyspnea and Fatigue will be assessed through Borg's perceived exertion scale
Dyspnea and Fatigue | Protocol 1: minute four; Protocol 2: minute eight
  Dyspnea and Fatigue will be assessed through Borg's perceived exertion scale
Dyspnea and Fatigue | Immediately after the session
  Dyspnea and Fatigue will be assessed through Borg's perceived exertion scale
Autonomic control | Baseline
  Autonomic control will be assessed through variability heart rate
Autonomic control | Up to 10 minutes after the session
  Autonomic control will be assessed through variability heart rate
Adverse events | Immediately after the session
  Occurrence of adverse events will be assessed through patient report
Adverse events | 24 hours after the session
  Occurrence of adverse events will be assessed through patient report
Adverse events | 48 hours after the session
  Occurrence of adverse events will be assessed through patient report
Adverse events | 72 hours after the session
  Occurrence of adverse events will be assessed through patient report

SECONDARY OUTCOMES:
Muscle damage | Baseline
  Assessed through the serum level of creatine kinase (CK)
Muscle damage | Immediately after the session
  Assessed through the serum level of creatine kinase (CK)
Muscle damage | 24 hours after the session
  Assessed through the serum level of creatine kinase (CK)
Muscle damage | 48 hours after the session
  Assessed through the serum level of creatine kinase (CK)
Muscle damage | 72 hours after the session
  Assessed through the serum level of creatine kinase (CK)
Muscle fatigue | Baseline
  Assessed through the serum lactate level
Muscle fatigue | Immediately after the session
  Assessed through the serum lactate level
Muscle fatigue | 3 minutes after the session
  Assessed through the serum lactate level
Muscle fatigue | 6 minutes after the session
  Assessed through the serum lactate level
Delayed onset muscle pain | Baseline
  Assessed by visual numerical scale, ranging from 0 to 10, where 0 indicates no pain and 10 indicates maximum pain.
Delayed onset muscle pain | Immediately after the session
  Assessed by visual numerical scale
Delayed onset muscle pain | 24 hours after the session
  Assessed by visual numerical scale
Delayed onset muscle pain | 48 hours after the session
  Assessed by visual numerical scale
Delayed onset muscle pain | 72 hours after the session
  Assessed by visual numerical scale
Peripheral muscle strength | Baseline
  Assessed by dynamometry
Peripheral muscle strength | Up to 40 minutes after the session
  Assessed by dynamometry

CONTACTS AND LOCATIONS:
Overall Officials: Jociane Schardong, Principal Investigator — Federal University of Health Sciences of Porto Alegre
Locations (1):
- Federal University of Health Sciences of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No